CLINICAL TRIAL: NCT03579407
Title: Traditional Open Ended Trocar vs. Fenestrated Blunt Trocar in Bone Marrow Aspirate for Osteoarthritis: A Randomized Controlled Trial
Brief Title: Open Ended Trocar vs. Fenestrated Blunt Trocar in Bone Marrow Aspirate for Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID limitations and staff changes
Sponsor: Advanced Orthopaedic Specialists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: bmacneedle
Record Dates: First submitted 2018-05-21; First posted 2018-07-06 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; cell therapy; stem cells; needle; bone marrow aspiration
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Traditional Open Ended Trocar (Active Comparator): Patients will undergo bone marrow aspiration using the Jamshidi bone marrow aspiration needle. This needle is the traditional trocar with an open end. 50-60 mL will be collected and concentrated with a centrifuge.
  Interventions: Procedure: BMA cell therapy injection
- Fenestrated Blunt Trocar (Experimental): Patients will undergo bone marrow aspiration using the Marrow Cellution bone marrow aspiration needle. This needle has several fenestrations along the trocar through which the bone marrow is aspirated. Approximately 8-10 mL of high concentrate bone marrow will be collected, which will not be concentrated.
  Interventions: Procedure: BMA cell therapy injection

INTERVENTIONS:
Procedure: BMA cell therapy injection — The bone marrow aspirate will be injected into the affected knee joint.

SUMMARY:
Osteoarthritis (OA) is a leading cause of disability around the world. The aging population is only further increasing its prevalence. Moreover, increasing rates of obesity, as well as increasing athletic participation, is leading to patients developing OA at younger ages. Although total joint replacement is effective for alleviating the effects of OA for many patients, it is less beneficial for younger patients given the resultant reduced mobility and the ~15 year life of a total joint replacement. Therefore, new options are needed for OA.

One such option is bone marrow aspirate concentrate (BMAC) injection into the diseased joint. Several recent studies have shown significant symptomatic improvement from this therapy. Now, efforts are needed to better understand how to optimize this therapy, as numerous variables are involved, including: the volume of aspirate, adjuvant, aspiration location or locations, anesthetic, etc. Additionally, several FDA-approved needles are available for the aspiration step. Thus, the purpose of this study is to compare two different styles of FDA-approved needles--an open-ended trocar vs. a fenestrated blunt trocar--with respect to clinical outcomes, cell counts, and colony forming units.

In addition to the comparison arms, taking these two groups together, this study will serve as prospective case series of 30 patients undergoing BMAC injection for knee osteoarthritis without a platelet-rich plasma (PRP) or any other adjuvant/carrier.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-79
* Patients have tried at least 6 weeks of conservative therapy including: activity modification, weight loss, brace, NSAIDs, corticosteroid injection
* Radiographically confirmed Kellgren-Lawrence I-III OA (no bone-on-bone)
* Patients can provide written informed consent

Exclusion Criteria:

* Clinically and radiologically confirmed anterior/posterior cruciate ligament deficiencies
* History of meniscal injury other than degenerative meniscal tears
* Presence of a degenerative meniscal tear causing mechanical symptoms such as locking, buckling, or give-way
* Major mechanical axis deviation of more than 50% into either compartment (varus or valgus)
* Intra-articular injection to affected knee within 3 months of intra-articular BMA injection or HA within 6 months
* Body mass index of 35 or more; 18.5 or less (malnourished)
* Active infection
* Ongoing infectious diseases, including HIV and hepatitis
* Clinically significant diabetes, cardiovascular, hepatic, or renal disease
* Active malignancy, undergoing treatment, has undergone treatment, or has decline treatment
* Use of anti-inflammatory medications, including herbal therapies, within 7 days of BMA
* Use of anti-rheumatic medications, including methotrexate and other antimetabolites, within 3 months prior to study entry
* History of radiation therapy
* History of or current drug or alcohol use disorder
* Current cigarette smokers
* History of anemia, bleeding disorders, or inflammatory joint disease (rheumatoid arthritis, infectious arthritis, hemophilic arthropathy, Charcot's knee)
* History of metabolic bone disease (osteoporosis, osteomalacia, rickets, osteitis fibrosa cystica, Paget's disease of bone)
* Pregnant or currently breast-feeding
* Participation in a study of an experimental drug within 60 days of study entry

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Knee injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 1 week, 6 weeks, 6 months
  Will assess for change in patient reported outcome measure that assesses symptoms, stiffness, pain, function, and quality of life from pre-procedure to post-procedure.

SECONDARY OUTCOMES:
Change in Visual Analog Pain Scale (VAS) of affected knee | Baseline, 1 week, 6 weeks, 6 months
  Will assess for change in patient reported pain scale of the patient's affected/treated knee from pre-procedure to post-procedure.
Change in Lysholm Score | Baseline, 1 week, 6 weeks, 6 months
  Will assess for change in Lysholm patient reported outcome score from pre-procedure to post-procedure..
Change in Tegner Score | Baseline, 1 week, 6 weeks, 6 months
  Will assess for change in patient reported activity scale from pre-procedure to post-procedure.
Visual Analog Pain Scale (VAS) of aspiration site | Baseline (immediately after intervention), 1 week, 6 weeks, 6 months
  Will assess the patient reported pain scale of the patient's aspiration site immediately after intervention and changes at the various time points.

OTHER OUTCOMES:
Cell counts and colony forming units | 1x, immediately after intervention
  For each aspiration in the study, total nucleated cell counts and colony forming units will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Ylanon, M.D., Principal Investigator — Advanced Orthopaedic Specialists and University of Arkansas for Medical Sciences
Locations (1):
- Advanced Orthopaedic Specialists, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No